CLINICAL TRIAL: NCT07198308
Title: Association Between Blood Glucose Indicators and Heart Rate Variability in Non-diabetic Critically Ill Patients: a Single-center Prospective Study
Brief Title: Association Between Blood Glucose Indicators and Heart Rate Variability in Non-diabetic Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2025-586
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Heart rate variability (HRV) is a simple way to check how well the body's automatic nervous system is working. It does this by looking at how the heart rate changes in the electrocardiogram. HRV can be divided into time domain and frequency domain. Time domain indicators assess the tone of the autonomic nerves. Frequency domain indicators reflect the regulation of the sympathetic and parasympathetic nerves. An imbalance of the body's nervous system can be reflected by HRV. Stress hyperglycemia (SIH) is when your blood glucose levels go up because of an acute disease. This is usually related to the body's stress response, but if your blood glucose levels go up too much, it can lead to complications. A high blood sugar level caused by stress is common in intensive care units. There is a strong link between this and the death rate and how long patients stay there. There are lots of nerve endings in the pancreas. Nerve fibres control the way islet α/β cells work to keep the right amount of glucose in the blood. We know that the pancreatic nerve is important for controlling blood glucose levels, but we don't fully understand how it does this.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 99 years old
* Informed consent has been signed

Exclusion Criteria:

* Under 18 years old
* Diagnosed with diabetes either prior to or during hospitalization
* Missing HRV values
* Missing blood glucose and random insulin values

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who were hospitalized in the Intensive Care Unit of Zhongshan Hospital Affiliated to Fudan University after the start of the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between glucagon and HRV in non-diabetic critically ill patients | From enrollment to completion of indicator testing (within 24 hours)

SECONDARY OUTCOMES:
The correlation between blood glucose and random insulin levels and HRV in non-diabetic critically ill patients | From enrollment to completion of indicator testing (within 24 hours)